CLINICAL TRIAL: NCT05120687
Title: The Efficacy and Safety of Corticosteroid Combining Noncorticosteroid Systemic Immunomodulatory Therapy in VKH
Brief Title: Corticosteroid Combining Noncorticosteroid Systemic Immunomodulatory Therapy in VKH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, Lab of ocular immunology in Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2021NCSIT-VKH
Record Dates: First submitted 2021-10-15; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Vogt Koyanagi Harada Disease (VKH)
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome | interventions — Methotrexate; Adalimumab; Cyclophosphamide; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Corticosteroid group: Patients in corticosteroid group will receive systemic corticosteroid. In case of severe, the patients may receive methylprednisolone (no more than 1 gram/day) followed by gradual taper of oral prednisone.
- Corticosteroid + NCSIT group: Patients in corticosteroid + NCSIT group will receive systemic corticosteroids combined with Methotrexate or Adalimumab or other noncorticosteroid systemic immunomodulatory such as cyclophosphamide.
  Interventions: Drug: noncorticosteroid systemic immunomodulatory therapy (NCSIT)

INTERVENTIONS:
Drug: noncorticosteroid systemic immunomodulatory therapy (NCSIT) — Patients in corticosteroid + NCSIT group will receive systemic corticosteroids combined with Methotrexate 15mg/week or Adalimumab 40mg /2weeks or Mycophenolate Mofetil 1g/day or Cyclosporin 50mg-100mg/day or cyclophosphamide 10mg/kg on two consecutive days every 2 weeks.
  Other Names: Methotrexate; Adalimumab; cyclophosphamide; Cyclosporin; Mycophenolate Mofetil
  Groups: Corticosteroid + NCSIT group

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of corticosteroidcombining noncorticosteroid systemic immunomodulatory therapy (NCSIT) for the treatment of Vogt Koyanagi Harada disease (VKH).

DETAILED DESCRIPTION:
Vogt Koyanagi Harada disease (VKH) is a sort of autoimmune disease directed against uveal melanocytes, which is a common vision-threatening noninfectious uveitis in colored people. VKH patients given prednisone monotherapy are prone to relapse.

Noncorticosteroid systemic immunomodulatory therapy (NCSIT) demonstrated inflammation control and steroid-sparing effect in autoimmune diseases. Methotrexate as an antifolate metabolite has been widely used for its anti-inflammatory and immunomodulating properties. Adalimumab, humanized monoclonal anti-TNF-α antibody, have demonstrated the efficacy of noninfectious uveitis. Several randomized controlled trials have proved the efficacy and safety of NCSIT such as antimetabolite and biologics in non-infectious uveitis, while the optimal dose and treatment course remain unknown.

The investigators propose to explore the effect, safety and optimal dose of prednisone combining NCSIT in the treatment of VKH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis is based on Revised International Diagnostic Criteria (Read et al. 2001b).
* Age from 12 to 70 years old.
* Patients have no contraindication of prednisone and immunosuppressive therapy, as determined by the investigator based on the results of laboratory and physical examinations.
* Written informed consent is provided.

Exclusion Criteria:

* Patients with other ocular diseases or fundus diseases: diabetic retinopathy, neovascular/wet age-related macular degeneration
* History of renal or hepatic insufficiency, heart failure, systemic inflammatory disease or any other condition that, in the opinion of the investigator, would put the patients at risk by participating in the protocol.
* History of infectious disease like chronic or active hepatitis B infection, HIV infection, immunodeficiency syndrome, chronic recurring infections, or active tuberculosis.
* Female patients who were pregnant or considering becoming pregnant during the study.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: VKH patients treated at Zhongshan Ophthalmic Center between October 2021 and October 2025.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-10-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving corticosteroid-sparing effect | 6 months
  Corticosteroid-sparing effect is defined by the following: (1) less than or equal to 0.5+ anterior chamber cells, less than or equal to 0.5+ vitreous haze and no active retinal or choroidal lesions; (2) no more than 10 mg of oral prednisone per day; (3) all the above-mentioned description should be maintained over 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The aim of this study is to evaluate the efficacy and safety of prednisone combining noncorticosteroid systemic immunomodulatory therapy (NCSIT) for the treatment of Vogt Koyanagi Harada disease (VKH).